CLINICAL TRIAL: NCT01656707
Title: Adaptive Treatment for Adolescent Cannabis Use Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UConn Health (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PA08-263; R01DA030454 (NIH)
Record Dates: First submitted 2012-08-01; First posted 2012-08-03 (Estimated); Last update posted 2017-04-11 (Actual); Status verified 2017-04

CONDITIONS: Mental Disorders; Addictive Behaviors; Cannabis Use Disorder
Keywords: Adolescents; Substance Use Disorders
MeSH Terms: conditions — Mental Disorders; Behavior, Addictive; Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ACRA (Experimental): Ten weekly 60-minute sessions of Adolescent Community Reinforcement Approach (ACRA) will be provided as an Adaptive treatment condition.
  Interventions: Behavioral: ACRA
- Cognitive Behavioral Therapy (CBT) (Experimental): Ten weekly, 60-minute sessions of augmented individualized Cognitive Behavioral Therapy (CBT)will be provided as an Adaptive Treatment condition
  Interventions: Behavioral: CBT

INTERVENTIONS:
Behavioral: ACRA — Ten weekly,60-minute therapy sessions including six individual, two parent/guardian and two joint (individual and parent/guardian).
  Other Names: Adolescent Community Reinforcement Approach
  Arms: ACRA
Behavioral: CBT — 10 weekly, 60-minute sessions of augmented individualized CBT
  Other Names: Cogntive Behavioral Therapy
  Arms: Cognitive Behavioral Therapy (CBT)

SUMMARY:
The purpose of this study is to examine an Adaptive Treatment approach in order to improve outcomes of youth with Cannabis Use Disorders who are poor responders to treatment.

DETAILED DESCRIPTION:
The study will address the current contrasts in youth response to treatment, the problem of poor response to treatment and the prevention of relapse. Results from the study may support Adaptive Treatment as an efficacious approach for youth with Cannabis Use Disorder who are poor responders to treatment.

Poor responders fall into two categories, those who failed to achieve a negative drug urinalysis during the last session of the initial MET/CBT-7 treatment they attended, and those who either dropped out or were administratively discharged at any time during the initial MET/CBT-7 treatment.

ELIGIBILITY:
Inclusion Criteria:

* 13-18 years of age at the time of intake assessment
* Current diagnosis of DSM-IV Cannabis Abuse or Dependence
* Able to read and comprehend English at a 5th grade level
* Residence within 45 minutes drive from the UCHC Farmington treatment site
* Participant and a parent/legal guardian responsible for providing collateral information agree to sign an IRB approved consent form
* Participant and a parent/legal guardian responsible for providing collateral information agree to provide locator information
* The family is not planning to move from the area during the next six months

Exclusion Criteria:

* Meet criteria for dependence of any other substance of abuse other than nicotine or alcohol
* Report suicidal ideation with a plan, suicidal behavior, a plan to hurt oneself or other, or a history of self-injurious behavior all occurring in the last 30 days
* Meet a lifetime diagnosis of schizophrenia
* Has any current health (i.e. medical, psychiatric) condition that will compromise the participant's ability to regularly attend treatment
* Demonstrate an inability or unwillingness to provide locator information

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 172 (Actual)
Dates: Start 2011-09; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
1.) To evaluate the efficacy of AT for youth who have been defined as poor responders to an evidence-based practice intervention such as the initial MET/CBT-7. | one year
  Each participant will serve as his/her own control. The outcomes will include the T-ASI, T-ASI-P, and drug urinalyses.

SECONDARY OUTCOMES:
To assess outcomes as a function of mediator variables such as self-efficacy, coping skills, readiness to change, and environmental support (i.e., family and peer), within each of the AT interventions. | one year
  The secondary outcome measures will include the SCQ, CRI, PRQ, and SSQ.

CONTACTS AND LOCATIONS:
Overall Officials: Yifrah Kaminer, MD, MBA, Principal Investigator — UConn Health
Locations (1):
- University of Connecticut Health Center, Farmington, Connecticut, United States